CLINICAL TRIAL: NCT07377500
Title: Randomised Controlled Trial of Dialysate Cooling for the Preservation of Cognitive Function in People Receiving Haemodialysis
Brief Title: Dialysate Cooling for the Preservation of Cognitive Function in People Receiving Haemodialysis
Acronym: COOL HD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UHDB/2024/007; 345755 (Other: IRAS)
Record Dates: First submitted 2026-01-02; First posted 2026-01-30 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Haemodialysis; Kidney Failure
Keywords: DIALYSATE COOLING; KIDNEY FAILURE; HAEMODIALYSIS; COGNITIVE IMPAIRMENT
MeSH Terms: conditions — Renal Insufficiency; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessor of outcomes will be blinded to mitigate introduction of any potential bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard temperature dialysis (No Intervention): Dialysis with a dialysate temperature of 37 degrees
- Cooled dialysis (Active Comparator): Dialysis with a dialysate temperature of 0.5 degrees below body temperature.
  Interventions: Other: Dialysis cooling

INTERVENTIONS:
Other: Dialysis cooling — dialysis with a dialysate temperature of 0.5 degrees below body temperature for a period of one year.
  Arms: Cooled dialysis

SUMMARY:
When a person's kidneys are not working properly, they need a life-saving treatment called haemodialysis three times a week to filter the waste and extra fluids from the blood. 25 000 adults in the United Kingdom are currently having haemodialysis and unfortunately more than two-thirds of these people experience problems with thinking and memory, which may lead to dementia. These problems tend to worsen more rapidly than people who are not on haemodialysis. This decline in brain function can make it harder for people to do everyday tasks, increase their reliance on others, and lower their overall quality of life. It also raises the chances of needing hospital care and can shorten their lifespan.

One reason for this decline in thinking and memory could be the dialysis treatment itself. Research has shown that blood flow to the brain can drop during dialysis. If this happens regularly, it can harm the brain over time. Earlier studies found that cooling the dialysis fluid slightly (to 0.5°C below body temperature) helped people tolerate dialysis better and showed less brain damage on magnetic imaging brain scans (MRI) after a year, compared to those who had haemodialysis without cooling the dialysis fluid. However, the investigators still don't know if this brain protection translates into better thinking and memory for people on haemodialysis.

This study will see if cooling the dialysis fluid helps preserve thinking and memory function.

The investigators will invite participants at three hospitals with haemodialysis centres to take part. Those who agree will be randomly assigned to either standard dialysis or cooled dialysis. The investigators will assess participants' thinking and memory functions using special tests at the start of the study and again after a year. By comparing the results from both groups, the investigators hope to see if the cooled dialysis really helps protect brain.

DETAILED DESCRIPTION:
Cognitive impairment is increasingly recognised as a major problem in the 25,000 adults with kidney failure treated by haemodialysis in the United Kingdom. The onset of cognitive impairment happens early after starting haemodialysis, and has an accelerated course so that some degree of cognitive impairment is almost universal, and over two-thirds of patients have moderate to severe reductions on cognitive function testing. A systematic review and meta-analysis of cognition in people on haemodialysis found that their global cognitive function scores were 25% lower than the general population, particularly in the domains of working memory, attention, orientation and executive function. Furthermore, the one-year risk for developing multi-infarct dementia in people on haemodialysis is more than 7 times higher than the general population. Investigators previously studied brain white matter microstructure in haemodialysis patients using diffusion tensor magnetic resonance imaging (MRI) and demonstrated the presence of significant brain white matter damage in haemodialysis patients compared to aged-matched controls. The amount of brain white matter damage correlated with lower score in cognitive function tests. Cognitive impairment in people on haemodialysis is a major component of the frailty syndrome that is also common in this population and cognitive impairment leads to increased dependency, poor quality of life, and reduces the ability of patients to correctly take medications and follow other important aspects of treatment such as dietary and fluid restrictions. Furthermore, cognitive impairment is associated with reduced survival and higher rates of hospitalisation. This has a further detrimental impact on quality of life and results in additional costs to the health service.

Working memory is the ability to hold and manipulate information in mind in the short term, which enables completion of cognitive tasks. It is one of the executive functions and it is well established that these are predictors for ability to carry out activities of daily living such as managing medications and using transport, executive function test performance is a stronger predictor than general cognition for activities and is vital for decision making. Working memory has been suggested as a potential treatment target due to its importance as a predictor of function. Letter Number Sequencing (LNS) is a well established test for working memory, it is derived from the Wechsler Adult Intelligence Scale-III and Wechsler Adult Intelligence Scale-IV test batteries. The LNS has clear face validity as a test of working memory. The participant hears a sequence of letters and numbers and must sort them into separate sequences of letters and numbers in the correct order. Testing working memory using LNS in haemodialysis patients compared to healthy controls demonstrated significant impairment in haemodialysis patients' working memory. Currently there are no interventions proven to protect cognitive function in people on haemodialysis.

Although haemodialysis is life sustaining for those with kidney failure, it is increasingly recognised that the haemodynamic effects of the treatment itself have negative effects on the blood flow to various vascular beds. These effects manifest as intradialytic hypotension, myocardial hypoperfusion leading to myocardial stunning and brain hypoperfusion. Dialysate cooling was first tested as an intervention in the 1980s to reduce intradialytic hypotension. Since then, there has been a large body of evidence that demonstrated beneficial effect of dialysate cooling on blood pressure. Dialysate cooling has been found to improve the stability of blood pressure and reduce intradialytic hypotension, confirmed in two metanalyses.

In smaller studies, dialysate cooling has also been shown to protect against intradialytic cardiac dysfunction and ameliorate myocardial stunning. In a previous NIHR-funded randomised clinical trial, investigators tested the hypothesis that improved haemodynamic stability with dialysate cooling would reduce the development of ischaemic lesions in the brain as determined by diffusion tensor imaging (DTI) MRI. The investigators randomised 73 participants to dialysate cooling to 0.5○C below body temperature or standard dialysis at 37○C. After one-year the standard haemodialysis patients developed MRI changes consistent with ischemic brain injury (increased fractional anisotropy and reduced radial diffusivity), cooled dialysate improved hemodynamic tolerability, and this group were protected against the development of brain white matter changes. The trial was designed with DTI-MRI as the primary outcome measure, and this meant that the study was not powered or designed to assess the effect on cognitive function.

More recently, a large cluster randomised, registry-based pragmatic trial (MyTEMP) conducted in Canada failed to demonstrate that dialysate cooling led to survival benefit or reduction in major cardiovascular events. However methodological limitations, lack of granularity of patient-level data and absence of important patient-centred outcomes mean that these results do not address questions as to whether cooling the dialysate can improve patient-centred outcomes, including protection against the development of cognitive impairment.

OBJECTIVES AND OUTCOME MEASURES/ ENDPOINTS

Haemodialysis causes significant haemodynamic effects, often causing blood pressure drops and leading to reduced perfusion of cardiac and brain tissue. Subclinical ischaemic injury to the brain has therefore been suggested as a mechanism whereby haemodialysis may cause or accelerate cognitive impairment. Investigators previously conducted a randomised controlled trial that examined the effects of cooling the dialysis fluid to 0.5○C below body temperature, a simple intervention that reduces the fall in blood pressure during dialysis. Compared to standard dialysis with dialysis fluid temperature 37○C, this trial demonstrated that dialysate cooling preserved brain white matter microstructure as assessed by MRI. However, this trial was not designed to assess the effect of dialysate cooling on cognitive function and was not powered to do so. Building on this work, investigators now propose to test the hypothesis that cooling the dialysate to 0.5○C below body temperature preserves cognitive function in haemodialysis patients.

This randomised controlled trial will answer the important clinical question of whether dialysate cooling leads to preservation of cognitive function in people on haemodialysis, building upon our previous work showing this intervention preserves brain white matter structural integrity. This is an important patient centred outcome due to the impact of cognitive function on functional status and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* The participant is receiving maintenance in-centre haemodialysis
* Over 18 years of age at time of consent
* The participant is able and willing to provide written informed consent.

Exclusion Criteria:

* Participants with confirmed diagnosis of dementia.
* Participants who lack capacity to consent.
* Participants having dialysis less than three times a week.
* Pregnant participants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in working memory | One year from randomisation
  Change in working memory as measured by the Letter Number Sequencing (LNS) test after one year from randomisation.

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Eldehni, Principal Investigator — University of Nottingham
Locations (1):
- Royal Derby Hospital, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Selby NM, McIntyre CW. A systematic review of the clinical effects of reducing dialysate fluid temperature. Nephrol Dial Transplant. 2006;21(7):1883-98
- [Background] Sherman RA, Faustino EF, Bernholc AS, Eisinger RP. Effect of variations in dialysate temperature on blood pressure during hemodialysis. Am J Kidney Dis. 1984;4(1):66-8.
- [Background] Anazodo UC, Wong DY, Théberge J, Dacey M, Gomes J, Penny JD, et al. Hemodialysis-Related Acute Brain Injury Demonstrated by Application of Intradialytic Magnetic Resonance Imaging and Spectroscopy. J Am Soc Nephrol. 2023;34(6):1090-104
- [Background] Findlay MD, Dawson J, Dickie DA, Forbes KP, McGlynn D, Quinn T, et al. Investigating the Relationship between Cerebral Blood Flow and Cognitive Function in Hemodialysis Patients. J Am Soc Nephrol. 2019;30(1):147-58.
- [Background] Kanbay M, Ertuglu LA, Afsar B, Ozdogan E, Siriopol D, Covic A, Basile C, Ortiz A. An update review of intradialytic hypotension: concept, risk factors, clinical implications and management. Clin Kidney J. 2020 Jul 8;13(6):981-993. doi: 10.1093/ckj/sfaa078. eCollection 2020 Dec. PMID 33391741
- [Background] Assa S, Hummel YM, Voors AA, Kuipers J, Westerhuis R, de Jong PE, et al. Hemodialysis-induced regional left ventricular systolic dysfunction: prevalence, patient and dialysis treatment-related factors, and prognostic significance. Clin J Am Soc Nephrol. 2012;7(10):1615-23.
- [Background] Burton JO, Jefferies HJ, Selby NM, McIntyre CW. Hemodialysis-induced cardiac injury: determinants and associated outcomes. Clin J Am Soc Nephrol. 2009;4(5):914-20.
- [Background] McIntyre CW. Recurrent circulatory stress: the dark side of dialysis. Semin Dial. 2010;23(5):449-51
- [Background] Sánchez-Fernández MDM, Reyes Del Paso GA, Gil-Cunquero JM, Fernández-Serrano MJ. Executive function in end-stage renal disease: Acute effects of hemodialysis and associations with clinical factors. PLoS One. 2018;13(9):e0203424.
- [Background] Berger I, Wu S, Masson P, Kelly PJ, Duthie FA, Whiteley W, et al. Cognition in chronic kidney disease: a systematic review and meta-analysis. BMC Med. 2016;14(1):206.
- [Background] Brodski J, Rossell SL, Castle DJ, Tan EJ. A Systematic Review of Cognitive Impairments Associated With Kidney Failure in Adults Before Natural Age-Related Changes. J Int Neuropsychol Soc. 2019;25(1):101-14
- [Background] Gaubert F, Borg C, Chainay H. Decision-Making in Alzheimer's Disease: The Role of Working Memory and Executive Functions in the Iowa Gambling Task and in Tasks Inspired by Everyday Situations. Journal of Alzheimer's Disease. 2022;90:1793-815.
- [Background] McDougall GJ, Han A, Staggs VS, Johnson DK, McDowd JM. Predictors of instrumental activities of daily living in community-dwelling older adults. Archives of Psychiatric Nursing. 2019;33(5):43-50
- [Background] Baddeley A. Working memory. Science. 1992;255(5044):556-9.
- [Background] Joshi U, Subedi R, Poudel P, Ghimire PR, Panta S, Sigdel MR. Assessment of quality of life in patients undergoing hemodialysis using WHOQOL-BREF questionnaire: a multicenter study. Int J Nephrol Renovasc Dis. 2017;10:195-203.
- [Background] UK Renal Regisstry 23rd Annual Report, Chapter 5 - Adults on in-centre haemodialysis (ICHD) in the UK at the end of 2019 [Available from: https://ukkidney.org/sites/renal.org/files/23rd_UKRR_ANNUAL_REPORT_ICHD_Ch5_0.pdf
- [Background] Hain DJ. Cognitive function and adherence of older adults undergoing hemodialysis. Nephrol Nurs J. 2008;35(1):23-9.
- [Background] Kim EY, Lee YN. Coexisting with the Life of Patients with Hemodialysis: Qualitative Meta-Synthesis Study of Life of Caregivers of Patients with Hemodialysis. Int J Environ Res Public Health. 2022;19(4)
- [Background] Eldehni MT. Frailty, multimorbidity and sarcopaenia in haemodialysis patients. Curr Opin Nephrol Hypertens. 2022;31(6):560-5.
- [Background] Young HML, Ruddock N, Harrison M, Goodliffe S, Lightfoot CJ, Mayes J, et al. Living with frailty and haemodialysis: a qualitative study. BMC Nephrol. 2022;23(1):260.
- [Background] Eldehni MT, Odudu A, McIntyre CW. Brain white matter microstructure in end-stage kidney disease, cognitive impairment, and circulatory stress. Hemodial Int. 2019;23(3):356-65
- [Background] Fazekas G, Fazekas F, Schmidt R, Kapeller P, Offenbacher H, Krejs GJ. Brain MRI findings and cognitive impairment in patients undergoing chronic hemodialysis treatment. J Neurol Sci. 1995;134(1-2):83-8.
- [Background] Fukunishi I, Kitaoka T, Shirai T, Kino K, Kanematsu E, Sato Y. Psychiatric disorders among patients undergoing hemodialysis therapy. Nephron. 2002;91(2):344-7.
- [Background] O'Lone E, Connors M, Masson P, Wu S, Kelly PJ, Gillespie D, et al. Cognition in People With End-Stage Kidney Disease Treated With Hemodialysis: A Systematic Review and Meta-analysis. Am J Kidney Dis. 2016;67(6):925-35.
- [Background] Kavanagh NT, Schiller B, Saxena AB, Thomas IC, Kurella Tamura M. Prevalence and correlates of functional dependence among maintenance dialysis patients. Hemodial Int. 2015;19(4):593-600.
- [Background] Kurella Tamura M, Covinsky KE, Chertow GM, Yaffe K, Landefeld CS, McCulloch CE. Functional status of elderly adults before and after initiation of dialysis. N Engl J Med. 2009;361(16):1539-47